CLINICAL TRIAL: NCT05155384
Title: Comparison of Biopsychosocial and Conventional Approach in the Treatment of Bladder Pain Syndrome/Interstitial Cystitis
Brief Title: Biopsychosocial and Conventional Approach in Bladder Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ceren Gursen, Doc. Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA- 21109
Record Dates: First submitted 2021-12-10; First posted 2021-12-13 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
Keywords: chronic pain; pain neuroscience education; Bladder Pain Syndrome; Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial; Chronic Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- biopsychosocial model-based treatment (Experimental): Biopsychosocial model-based management will be applied including pain neuroscience education, functional exercises, and relaxation training.
  Interventions: Other: Pain Neuroscience Education; Other: Relaxation exercises; Other: Cognition target exercise
- Conventional physiotherapy (Active Comparator): Conventional physiotherapy will be applied including standard exercises and electrical stimulation.
  Interventions: Other: Pelvic floor stretching exercises; Device: Transcutaneous electrical nerve stimulation

INTERVENTIONS:
Other: Pain Neuroscience Education — main topics of pain neuroscience education; neurophysiology of the nervous system, protective mechanism of pain, acute pain formation and chronic pain, factors that increase/reduce pain, central sensitization mechanism, neuroplasticity and treatment strategies in chronic pain.
  Arms: biopsychosocial model-based treatment
Other: Relaxation exercises — Relaxation exercises are a training based on deep relaxation techniques and visual imagery. Relaxation exercises will be applied at the end of the training sessions.
  Arms: biopsychosocial model-based treatment
Other: Cognition target exercise — Cognition target exercises are a time-based approach that is not symptom-conditioned (not based on fatigue or pain). It includes functional and dynamic exercises.
  Arms: biopsychosocial model-based treatment
Other: Pelvic floor stretching exercises — Pelvic floor stretching exercises; consists of stretching exercises involving the pelvic floor muscles and surrounding group muscles (such as piriformis, hamstring, adductor group muscles and lumbar extensors).
  Arms: Conventional physiotherapy
Device: Transcutaneous electrical nerve stimulation — It will be used with superficial electrodes attached to the suprapubic region of the patients for 20 minutes in each session.
  Arms: Conventional physiotherapy

SUMMARY:
The aim of the present study is to compare the effects of biopsychosocial and conventional approach on symptom severity, pain parameters (pain intensity and pain cognitions), disability, psychological distress and quality of life in patients who are suffering from bladder pain syndrome/interstitial cystitis. The study is designed as a randomized clinical trial including two parallel arms.

Individuals who meet the inclusion criteria and agree to participate will be randomly assigned into one of the two research arms: biopsychosocial approach group or conventional approach group. A biopsychosocial approach, which is a holistic approach that includes pain neuroscience education, relaxation training and cognitive exercises, will be applied to the patients in the first research arm for the treatment of chronic pain symptoms. For the patients in the second research arm, a conventional approach including pelvic floor stretching exercises and Transcutaneous Electrical Nerve Stimulation (TENS) will be applied for the treatment of chronic pain complaints. Treatments will be lasted for a total of six weeks, with two sessions per week. Participants will be evaluated at the baseline (before treatments) and at the end of the 6th week (after treatments). In the evaluations, information about the demographic and physical characteristics, medical and surgical background, medications and lifestyle characteristics (water, tea, coffee, alcohol, cigarette consumption, the presence constipation and physical activity level) of the individuals will be recorded. For primary or secondary outcome measures, Interstitial Cystitis Symptom and Problem Index, Visual Analog Scale, Pain Catastrophizing Scale, Pain Self-Efficacy Questionnaire, 3-day voiding diary, Pain Disability Index, Hospital Anxiety and Depression Scale, and Short Form-36 will be used. The present study is planned to be carried out with a total of 60 individuals, 30 for each study group based on a sample size analysis.

After reaching required sample for the present study, in patients with bladder pain syndrome/interstitial cystitis, the effects of biopsychosocial and conventional approach on symptom and problem severity, pain parameters, disability, psychological status and quality of life will be analyzed using (2*2) two-way ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Bladder Pain Syndrome/Interstitial Cystitis
* with chronic symptoms (more than 6 months)
* Bladder pain severity in the last week should be at least 3/10 according to the Visual Analogue Scale (VAS)
* Stable medication schedule
* Individuals over the age of 18 (individuals over 65 years of age with a Mini Mental Test score ≥ 24) voluntarily to participate in the study will be included.

Exclusion Criteria:

* Acute disease state (with ongoing urinary tract infection, active vaginitis, active Herpes infection)
* Stones in the bladder, ureter, or urethra in the last 3 months
* Having an ulcer appearance on cystoscopy
* For women: during pregnancy and/or breastfeeding
* Previous history of urological and/or pelvic malignancy
* Congenital anomaly of the upper and/or lower urinary tract
* who have started a new drug treatment in the last 3 months, or undergoing implantation operation of neuromodulation devices
* Diagnosed with opioid dependence
* Neurogenic bladder dysfunction or concomitant neurologic conditions
* Not cooperating with assessment and/or treatment, and illiterate individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
severity of symptoms | change in severity of symptoms from baseline up to end of 6th week
  The Interstitial Cystitis Symptom and Problem Index will be used to assess the severity of symptoms. This scale consists of two separate parts as symptom and problem index, both of which are four questions. Participants will be asked to fill in both parts.

SECONDARY OUTCOMES:
severity of pain | change in severity of pain from baseline up to end of 6th week
  Pain severity will be evaluated with the Visual Analogue Scale (VAS). Considering the last week, the patients will be asked to mark the severity of pain on a 10-centimeter (cm) straight line, with the starting end as "no pain" and the ending end as "unbearable pain". It will be calculated in cm by measuring the starting tip and the part marked by the patient.
Pain cognitions | change in pain cognitions from baseline up to end of 6th week
  Pain Catastrophizing Scale and Pain Self-Efficacy Questionnaire will be used to assess individuals' cognitions about pain (catastrophizing and self-efficacy).
urinary symptoms | change in urinary symptoms from baseline up to end of 6th week
  A 3-day voiding diary will be used to evaluate Urinary Symptoms. On this chart, they are asked to record the time they urinate, the amount of urine, the presence of urinary incontinence, the amount and type of fluid consumed.
severity of disability | change in severity of disability from baseline up to end of 6th week
  The Pain Disability Index will be used to question the impact of individuals' daily life due to their pain and the resulting disability.
psychological distress | change in psychological distress from baseline up to end of 6th week
  The Hospital Anxiety and Depression Scale will be used to evaluate the psychological distress of individuals. The questionnaire has two sub-dimensions, depression and anxiety.
quality of life of the patients | change in quality of life from baseline up to end of 6th week
  Quality of Life will be assessed using the SF-36 scale. Short Form-36 will be used for evaluations. This questionnaire consists of eight different sub-parameters (physical function, physical role difficulty, general health status, pain status, energy/fatigue, social function, emotional role difficulty, and emotional well-being).

CONTACTS AND LOCATIONS:
Overall Officials: Ceren Gürşen, PhD, Principal Investigator — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara
  - Hacettepe University, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Leary MP, Sant GR, Fowler FJ Jr, Whitmore KE, Spolarich-Kroll J. The interstitial cystitis symptom index and problem index. Urology. 1997 May;49(5A Suppl):58-63. doi: 10.1016/s0090-4295(99)80333-1. PMID 9146003
- [Background] Von Korff M, Jensen MP, Karoly P. Assessing global pain severity by self-report in clinical and health services research. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3140-51. doi: 10.1097/00007632-200012150-00009. No abstract available. PMID 11124730
- [Background] Suren M, Okan I, Gokbakan AM, Kaya Z, Erkorkmaz U, Arici S, Karaman S, Kahveci M. Factors associated with the pain catastrophizing scale and validation in a sample of the Turkish population. Turk J Med Sci. 2014;44(1):104-8. doi: 10.3906/sag-1206-67. PMID 25558568
- [Background] Nicholas MK. The pain self-efficacy questionnaire: Taking pain into account. Eur J Pain. 2007 Feb;11(2):153-63. doi: 10.1016/j.ejpain.2005.12.008. Epub 2006 Jan 30. PMID 16446108
- [Background] Pollard CA. Preliminary validity study of the pain disability index. Percept Mot Skills. 1984 Dec;59(3):974. doi: 10.2466/pms.1984.59.3.974. No abstract available. PMID 6240632
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Ware JE Jr. SF-36 health survey update. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3130-9. doi: 10.1097/00007632-200012150-00008. No abstract available. PMID 11124729
- [Background] Fitzgerald MP, Anderson RU, Potts J, Payne CK, Peters KM, Clemens JQ, Kotarinos R, Fraser L, Cosby A, Fortman C, Neville C, Badillo S, Odabachian L, Sanfield A, O'Dougherty B, Halle-Podell R, Cen L, Chuai S, Landis JR, Mickelberg K, Barrell T, Kusek JW, Nyberg LM; Urological Pelvic Pain Collaborative Research Network. Randomized multicenter feasibility trial of myofascial physical therapy for the treatment of urological chronic pelvic pain syndromes. J Urol. 2013 Jan;189(1 Suppl):S75-85. doi: 10.1016/j.juro.2012.11.018. PMID 23234638